CLINICAL TRIAL: NCT01951976
Title: Evaluating Yoga for Aromatase Inhibitor-associated Joint Pain in Women With Breast Cancer: A Pilot Study
Brief Title: Yoga for Aromatase Inhibitor-associated Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-17592
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: breast; carcinoma; stage 0-III breast cancer; post-menopausal; aromatase inhibitor (AI); joint pain; AI-associated joint pain
MeSH Terms: conditions — Breast Neoplasms; Carcinoma; Arthralgia | interventions — Surveys and Questionnaires; Yoga; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Condition (Experimental): Questionnaires and yoga classes.
  Group will attend a series of 90-minute yoga classes twice a week for 12 weeks.
  Interventions: Other: Questionnaires; Other: Yoga Classes

INTERVENTIONS:
Other: Questionnaires — Participants will be asked to complete a set of questionnaires about their health and well-being on two occasions (baseline and follow-up). Each set of questionnaires will take about 45 minutes to complete.
Other: Yoga Classes — Iyengar yoga is a traditional form of Hatha yoga that has been used previously to address quality of life issues in women with breast cancer. Iyengar yoga classes for 90 minutes twice per week for 12 weeks (total of 24 classes).
  Other Names: Iyengar yoga; yoga; exercise; Hatha yoga

SUMMARY:
The purpose of this study is to determine whether it might be practical and useful to investigate the effectiveness of yoga classes in relieving joint pain associated with the use of a class of medications known as aromatase inhibitors.

DETAILED DESCRIPTION:
The study uses a single-arm design. All study participants will be assigned to an intervention condition in which they participate in group Iyengar yoga classes for 90 minutes twice per week for 12 weeks (total of 24 classes). Study outcomes are assessed: 1) following recruitment but prior to the first yoga class; and 2) within two weeks post-intervention (follow-up). Additionally, a brief assessment of pain will be conducted four weeks and eight weeks after the start of yoga classes.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with stage 0-III breast cancer
* Have completed local and/or adjuvant breast cancer therapy (with the exception of hormonal therapy) at least one month previously
* Are post-menopausal defined as defined as no menses in the past 12 months
* Are currently prescribed an aromatase inhibitor (AI) medication (anastrozole, letrozole, or exemestane) by a Moffitt-affiliated physician
* Report joint pain that started or worsened after initiation of AI medication
* Report worst pain score > 4 in the preceding week on an 11-point (0-10) numeric rating scale

Exclusion Criteria:

* Have been diagnosed with another form of cancer (except nonmelanoma skin cancer) in the last five years
* Have uncontrolled cardiac disease, pulmonary disease, or infectious disease
* Have physical symptoms or conditions that could make yoga unsafe (i.e., neck injuries, dizziness, shortness of breath, chest pain, or severe nausea)
* Have a body mass index (BMI) > 40 kg/m^2 (based on difficulties severly obese individuals may have with engaging in Iyengar yoga poses)
* Have joint pain attributed to inflammatory arthritic conditions (i.e., rheumatoid arthritis, gout, pseudo-gout) per medical record or patient history
* Had surgery within the past 3 months
* Had injections of medication within the last 3 months to joint(s) currently painful
* Are currently using corticosteroids or opioid medications
* Are currently attending yoga classes
* Do not speak or read standard English
* Are scheduled or are planning to discontinue AI medication in the next 16 weeks
* Do not have sufficient access to the Internet to complete study assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rate of Study Enrollment | 24 months
  Acceptability of the proposed study to potential participants. The study will be considered acceptable if 50% or more of eligible participants agree to participate.
Rate of Study Completion | Up to 24 weeks per participant
  Feasibility of the proposed study assessment and intervention methods. The study methods will be considered feasible if 70% or more of consented participants complete both the baseline and follow-up assessments and attend an average of 70% or more of scheduled yoga classes.

SECONDARY OUTCOMES:
Occurrence of Reduced Pain Severity | Up to 24 weeks per participant
  Potential efficacy of the intervention in relieving AI medication-associated joint pain. The intervention will be considered potentially efficacious in relieving AI medication-associated joint pain if comparisons of pre- and post-intervention means for one or more measures of pain severity yield an effect size >/= 0.3 consistent with pain reduction.
Occurrence of Relief from Other Side Effects | Up to 24 weeks per participant
  Potential efficacy of the intervention in relieving other reported side effects of AI medication (i.e., fatigue, hot flashes, sleep problems, and depressive symptoms). The intervention will be considered potentially efficacious in relieving other known side effects if comparisons of pre- and post-intervention means yield an effect size >/= 0.3 consistent with side effect reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Jacobsen, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States